CLINICAL TRIAL: NCT06830967
Title: Virtual Prehabilitation for Patients Undergoing Abdominal Aortic Aneurysm Repair
Acronym: VPAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Samuel Jessula, Assistant Professor in Surgery, Division of Vascular Surgery, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68360
Record Dates: First submitted 2025-01-29; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Aortic Aneurysm; Prehabilitation; AAA - Abdominal Aortic Aneurysm
Keywords: AAA; prehabilitation; abdominal aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Preoperative Exercise; Exercise Therapy; Psychosocial Intervention; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prehabilitation arm (Experimental): Participants in the intervention arm will receive a prehabilitation bundle between the time of diagnosis of abdominal aortic aneurysm and open surgical repair. The prehabilitation bundle will consist of 5 main interventions: exercise therapy; smoking cessation counseling and pharmacotherapy; nutritional counseling; psychological readiness planning and patient education. Exercise therapy will consist of 6 weeks of prescribed moderate exercise coordinated remotely through the physiotherapy. Smoking cessation will consist of motivational interview with adjunctive pharmacotherapy prescribed as required. Nutritional assessment will be remotely coordinated with a certified dietician and psychological readiness and patient education will consist of 2 1 hour sessions with a counselor.
  Interventions: Other: Prehabilitation; Behavioral: Exercise therapy; Behavioral: Smoking cessation counselling; Behavioral: Nutritional counselling; Behavioral: Psychological intervention; Behavioral: Patient Education

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation will consist of exercise therapy, smoking cessation, nutritional counselling, psychological intervention and patient education.
Behavioral: Exercise therapy — Exercise therapy will consist of tailored 6-week prescribed exercise program consisting of 150-minutes of moderate-vigorous exercise weekly based on patient-to-patient resource availability (eg. neighborhood walk, body-weight exercises). It will target moderate intensity (11-13 on the Borg Rating of perceived exertion scale) and will be adjusted throughout the program as required. It will target aerobic, strength and inspiratory muscle training (IMT). Participants will receive a logbook where the exercise specialist will prescribe the intensity, type, time, and frequency of aerobic, strength and IMT exercises. Each time the participant performs the prescribed home-based exercises they will register their activity in the logbook provided. Exercise specialist will review the logbook every week and will adjust the home-based exercise plan accordingly to ensure both safety and exercise progression.
Behavioral: Smoking cessation counselling — Smoking cessation will be provided through motivational interviewing with a counselor who will assess participant's smoking status, willingness and readiness to quit and provide prescriptions for nicotine replacement therapy in combination with non-nicotinic pharmacotherapy (Varenicline, Buprorprion) as appropriate
Behavioral: Nutritional counselling — Nutritional counseling will be provided through consultation with a registered dietician. Participants will be educated on correct portion sizes, building a balanced plate, learning sources and importance of protein, importance of timing and spacing of meals, along with practicing mindful eating. Promotion and encouragement of dietary changes to ensure balanced intake with adequate protein, weight management, and the regulation of blood glucose will be discussed. Possible barriers to attain the proposed dietary changes and ways to overcome them will also be discussed along with the importance of perioperative nutrition. Based on estimated habitual protein intake, participants will receive a tailored dietary advice aiming a total protein intake of 1,2-1,5g /kg daily, unless contraindicated. Also, participants will be recommended to evenly 'spread' their protein intake over 3 meals with a minimum of 25-30 gram of protein/ meal.
Behavioral: Psychological intervention — Participants will receive one hourly session of psychological intervention called "surgical stress tolerance training" with a trained counselor. In this session the psychosocial specialist will address the patient's anxieties, coping strategies, and post-operative expectations, with the goal of optimizing psychological well-being and ways of coping with surgery. The importance of the patient's active participation in the preparation for surgery and healing process will also be discussed. All participants will be given instructions on relaxation and deep breathing techniques.
Behavioral: Patient Education — Patient education will be provided through virtual consultations with a vascular surgery nurse practitioner. These consultations will describe to the patient their journey pre and post-operatively, what to expect and what they are likely to experience, both physically and emotionally. These consultations will also ensure participants have a support person at home available for supervision during prehabilitation and available during their recovery. Additionally, they will ensure that their home is organized for their discharge from hospital and if required, an occupational therapy home consultation may be organized.

SUMMARY:
The time between diagnosis and operative intervention represents an untapped opportunity to optimize patient readiness for surgery and augment their function prior to undergoing a physiological stress, rather than purely recovering post-operatively. Vascular surgery patients are frail and primed to benefit from such interventions and upcoming surgery is a strong motivator for behavioral change. In this proposal, the investigators outline our vision for a prehabilitation program for patients undergoing elective open aortic aneurysm repair (AAA).

Participants scheduled to undergo AAA repair would receive, in addition to standard of care, 5 main interventions: exercise therapy; smoking cessation counseling and pharmacotherapy; nutritional counseling; psychological readiness planning and patient education. Exercise therapy will consist of 6 weeks of moderate exercise coordinated remotely through the cardiology rehabilitation program, whereas all other interventions will be consultations through videoconferencing or phone interactions. Outcomes of interest include morbidity, mortality, predictors of completion of program, exercise function and quality of life.

This study is a pilot feasibility project and the first step in the creation of a long-term program that will improve patient clinical outcomes, exercise capacity quality of life and hopefully become an model for prehabilitation for other institutions across the country and raise the standard of care for vascular surgery patients.

DETAILED DESCRIPTION:
The time between diagnosis and operative intervention represents an untapped opportunity to optimize patient readiness for surgery and augment their function prior to undergoing a physiological stress, rather than purely recovering post-operatively. Vascular surgery patients are frail and primed to benefit from such interventions and upcoming surgery is a strong motivator for behavioral change. In this proposal, the investigators outline our vision for a prehabilitation program for patients undergoing elective open aortic aneurysm repair (AAA).

Participants scheduled to undergo AAA repair would receive, in addition to standard of care, 5 main interventions: exercise therapy; smoking cessation counseling and pharmacotherapy; nutritional counseling; psychological readiness planning and patient education. Exercise therapy will consist of 6 weeks of prescribed moderate exercise coordinated remotely through the physiotherapy. Smoking cessation will consist of motivational interview with adjunctive pharmacotherapy prescribed as required. Nutritional assessment will be remotely coordinated with a certified dietician and psychological readiness and patient education will consist of 2 1 hour sessions with a counselor. Outcomes of interest include morbidity, mortality, predictors of completion of program, exercise function and quality of life.

This study is a pilot feasibility project and the first step in the creation of a long-term program that will improve patient clinical outcomes, exercise capacity quality of life and hopefully become an model for prehabilitation for other institutions across the country and raise the standard of care for vascular surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 50 years of age awaiting elective open AAA repair with AAA diameter ≤6.9cm at the Halifax Infirmary Hospital between January 2025-December 2025. Participants must have the ability to give individual informed consent.

Exclusion Criteria:

* Participants undergoing thoracic, thoracoabdominal and/or perivisceral AAA repair.
* Participants with ruptured or symptomatic AAA.
* Participants with AAA maximal diameter ≥7cm.
* Physical inability to exercise: severe osteoarthritis, musculoskeletal or neurological impairment that precludes exercise.
* Contraindication to exercise: rest systolic blood pressure ≥ 180 mmHg and/or diastolic ≥ 100 mmHg, uncontrolled atrial or ventricular arrythmias or proven exercise induced arrhythmias, unstable angina, unstable or acute heart failure, severe symptomatic valvular stenosis, dynamic left ventricular outflow tract obstruction or other comorbidities that imply clinical instability.
* Inability to have a support person present during exercise therapy.
* Cognitive impairment that would impede understanding of study procedures or informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications measured by the Comprehensive Complication Index (CCI) | CCI will be measured from admission to 6 weeks postoperatively
  The CCI was developed to address some of the limitations of traditional surgical morbidity reporting, such as only reporting the most severe complication or only picking the most common types of complications. It is scored on a true linear interval scale from 0-100 and incorporates the totality of all complications and their severity experienced by a patient

SECONDARY OUTCOMES:
Change in aerobic function | Measured at baseline, preoperatively and 6 weeks postoperatively
  Change in 6 minute walk test. The 6 minute walk test is the maximum distance walked within a 6 minute time frame.
Physical activity | Measured at baseline, preoperatively and 6 weeks postoperatively
  Measured by the Yale physical activity survey (YPAS). The YPAS has 2 sections that provide 3 summary indices and a seasonal adjustment score, all of which are calculated as a recall of physical activity in a typical week in the past month. The range is 0-142, with higher scores suggesting higher physical activity.
Quality of life | Measured at baseline, preoperatively and 6 weeks postoperatively
  The SF 36 measures eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions via survey. The SF 36 range is 0-100, with higher scores indicting higher quality of life.
Anxiety | Measured at baseline, preoperatively and 6 weeks postoperatively
  Anxiety measured by the Hospital Anxiety and Depression questionnaire (HADS) 0 (no anxiety)- 21 (maximal anxiety).
Compliance | Measured from baseline to preoperatively
  Compliance to the different components of the intervention, measured by attendance to supervised sessions (%), adherence to nutritional counseling and supplementation (%), adherence to home-based exercise (%) and adherence to the psychosocial sessions (%)
ICU Length of stay | From admission to 6 weeks postoperatively
  Intensive Care Unit length of stay
Hospital length of stay | From admission to 6 weeks postoperatively
  Days from admission to discharge from the hospital
Reinterventions | From admission to 6 weeks postoperatively
  Need for surgical reintervention due to surgical complications
Readmission | at 6 weeks and at 1 year postoperatively
  Readmission to the hospital
Emergency Room visits | at 6 weeks and at 1 year postoperatively
  Visits to the emergency room with or without admission to the hospita
Mortality | From admission to 1 year post operatively.
  Mortality within 1 year of surgery.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect patient privacy.